CLINICAL TRIAL: NCT06942715
Title: Applied Implementation Research for Clean Cooking in Cambodia: Equity, Exposure, Costs, and Benefits of Induction Stove Interventions
Brief Title: Applied Implementation Research for Clean Cooking in Cambodia
Acronym: AIR-C3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Matthew Freeman, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00007929; 1R01ES035395-01A1 (NIH); 2025P013174 (Other: Emory IRB)
Record Dates: First submitted 2025-03-24; First posted 2025-04-24 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Exposure to Environmental Pollution; Exposure to Household Air Pollution
Keywords: Cooking methods; Induction stoves

STUDY DESIGN:
Intervention Model Description: Hybrid type II cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- "Standard" implementation delivery (Experimental): The intervention will be promoted through a combination of (1) digital outreach and (2) community-centered demand generation. This includes:
  1. Low-touch awareness raising through geo-targeted social media promotion.
  2. In-person, village-level promotion through community engagement and local communication channels to raise awareness and build trust
  Interventions: Other: Electric Induction Cookstoves
- "Standard Plus" implementation delivery (Experimental): The intervention will be promoted through a combination of (1) digital outreach and (2) community-centered demand generation, paired with (3) stove subsidies. This includes:
  1. Low-touch awareness raising through geo-targeted social media promotion.
  2. In-person, village-level promotion through community engagement and local communication channels to raise awareness and build trust.
  3. Lower-value, untargeted stove subsidy for all households and a higher-value, targeted subsidy for low-income households to improve affordability and access.
  Interventions: Other: Electric Induction Cookstoves
- "Enhanced" implementation delivery (Experimental): The intervention will be promoted through a combination of (1) digital outreach, (2) community-centered demand generation, and (3) direct sales. This includes:
  1. Low-touch awareness raising through geo-targeted social media promotion.
  2. In-person, village-level promotion through community engagement and local communication channels to raise awareness and build trust.
  3. Door-to-door and group-based direct sales efforts to engage customers, demonstrate products, and facilitate purchases.
  Interventions: Other: Electric Induction Cookstoves
- "Enhanced Plus" implementation delivery (Experimental): The intervention will be promoted through a combination of (1) digital outreach, (2) community-centered demand generation, and (3) direct sales, paired with (4) stove subsidies. This includes:
  1. Low-touch awareness raising through geo-targeted social media promotion.
  2. In-person, village-level promotion through community engagement and local communication channels to raise awareness and build trust.
  3. Door-to-door and group-based direct sales efforts to engage customers, demonstrate products, and facilitate purchases.
  4. Lower-value, untargeted stove subsidy for all households and a higher-value, targeted subsidy for low-income households to improve affordability and access
  Interventions: Other: Electric Induction Cookstoves
- "Reference" implementation delivery (Active Comparator): The intervention will be promoted through only digital outreach, using low-touch awareness raising through geo-targeted social media promotion.
  Interventions: Other: Electric Induction Cookstoves

INTERVENTIONS:
Other: Electric Induction Cookstoves — The intervention consists of high-quality, locally available electric induction cookstoves with one or two burners, each equipped with cloud-connected data loggers, and includes compatible cookware.

SUMMARY:
The goal of this study is to learn how to help families in Cambodia switch to using electric induction stoves instead of traditional stoves that burn wood or charcoal. The study will also look at whether this switch is safe, affordable, and sustainable over time.

The main questions researchers want to answer are:

* What strategies work best to encourage families to use induction stoves regularly and stop using traditional cooking methods?
* Does switching to induction cooking reduce household air pollution for primary cooks?
* What are the costs and benefits of these strategies?

To answer these questions, researchers will compare four different strategies across 62 peri-urban villages in Cambodia. They will use data loggers to track when families use induction stoves or traditional stoves, and measure air pollution levels in the home before and after families receive induction stoves.

Participants will:

* Receive an electric induction stove and support based on their group's strategy
* Have their stove use tracked through special devices
* Take part in air pollution measurements in their homes
* Share information about their cooking habits and experiences

DETAILED DESCRIPTION:
Around 3 billion people worldwide cook using biomass fuels like wood, charcoal, and animal dung, which creates household air pollution responsible for about 2.3 million premature deaths each year from diseases such as heart disease, respiratory illnesses, diabetes, and cancer. Previous efforts to clean up biomass fuel burning have not sufficiently reduced air pollution or replaced traditional stoves, leading researchers to explore even cleaner alternatives like electric induction cooking.

This study evaluates whether electric induction stoves can effectively lower household air pollution in Cambodia. Using a rigorous, multi-year, cluster-randomized trial in 62 peri-urban villages, the study will:

* Develop and test different strategies (such as direct sales, subsidies, and community promotion) to encourage the purchase and regular use of induction stoves.
* Measure stove usage with cloud-connected data loggers that record cooking times and energy consumption.
* Collect household air pollution data and conduct surveys and interviews with approximately 3,100 households, with a focus on primary cooks.

The study also includes a comprehensive cost-effectiveness analysis to understand the benefits in terms of health, environmental impact, time savings, and equity, especially for women and girls who primarily prepare food. By using established frameworks like (RE-AIM) and Consolidated Framework for Implementation Research (CFIR), the research aims to build a strong evidence base to support the scale-up of clean cooking interventions in Cambodia and other low- and middle-income settings.

ELIGIBILITY:
Inclusion Criteria:

- A household must:

* Provide consent to participate in our study, with at least one adult household member who identifies as the primary cook consenting to serve as the study participant
* Resides in village selected for implementation
* Household has electricity access
* Household does not already use electricity-based induction cooking technology

Exclusion Criteria:

* Household members currently smoke cigarettes or other tobacco products
* Plans to move permanently outside the study area in the next 12 months
* The primary cook prepares food and/or drink for commercial sale

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6150 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Induction stove purchase: Proportion of eligible households that purchase an induction stove, based on study and sales records | 12 months, at the end of intervention completion
  This outcome will assess the proportion of eligible households that purchase an induction stove during the intervention period. Purchase data will be tracked through verified sales receipts linked to household study IDs. The outcome will be calculated as the number of participating households with a confirmed induction stove purchased divided by the total number of households in the enrolled community. Results will be reported overall and stratified by household income status.
Induction stove use: Number of daily cooking events | Up to 30 months following stove purchase
  This outcome will assess the intensity of induction stove use derived from built-in stove usage data loggers installed on all induction stoves sold to participants. All participating households that purchase an induction stove and consent to follow-up monitoring will have induction stove usage recorded up to 30 months following stove purchase. These devices log time-of-use for each induction surface/burner and energy used by the stove during cooking. This metric will count the number of daily cooking events.
Induction stove use: Duration of daily cooking | Up to 30 months following stove purchase
  This outcome will assess the intensity of induction stove use derived from built-in stove usage data loggers installed on all induction stoves sold to participants. All participating households that purchase an induction stove and consent to follow-up monitoring will have induction stove usage recorded up to 30 months following stove purchase. These devices log time-of-use for each induction surface/burner and energy used by the stove during cooking. This metric will evaluate the duration of stove use per day
Induction stove use: Daily electricity consumption of cooking events | Up to 30 months following stove purchase
  This outcome will assess the intensity of induction stove use derived from built-in stove usage data loggers installed on all induction stoves sold to participants. All participating households that purchase an induction stove and consent to follow-up monitoring will have induction stove usage recorded up to 30 months following stove purchase. These devices log time-of-use for each induction surface/burner and energy used by the stove during cooking. This metric will evaluate the amount of energy used per day by the induction stove unit: (electricity consumption in kWh)

SECONDARY OUTCOMES:
Biomass stove disuse: Proportion of days with no biomass stove use among households that purchased an induction stove | Daily, over a 1-week period following stove purchase
  This outcome will measure how many households stop using traditional biomass stoves after purchasing an induction stove. Participating households that consent to follow-up will have biomass stove use monitored for 7 days, between 6-8 weeks after purchase. Monitoring will use Geocene Dots-thermocouple-based temperature loggers that record stove temperatures and transmit data via Bluetooth to mobile devices, which sync to a central server. A validated algorithm will convert temperature data into daily usage metrics (number and duration of cooking events). The outcome will be reported as the proportion of days with no biomass stove use. Data will be aggregated across up to 2,400 households, with results stratified by income status.
Determinants: Induction stove purchase and use determinants | 30 months
  This outcome will assess household- and individual-level determinants associated with the purchase and use of induction stoves and continued use of biomass stoves. Structured survey data will be collected from all enrolled households at baseline and again at endline. Data will be analyzed to identify key factors associated with induction stove purchase, frequency and intensity of induction stove use, and continued use of biomass stoves. Results will be reported overall and stratified by household income status
Personal exposure: Changes in personal 24-hour exposure to PM2.5 among primary cooks, measured before and after the intervention | 30 months
  This outcome will assess changes in 24-hour personal exposure to fine particulate matter (PM2.5) among primary household cooks following the purchase of induction stoves. PM2.5 exposure will be measured using wearable personal exposure monitors placed in the breathing zone of the primary cook for a continuous 24-hour period. Measurements will be collected from approximately 600 households at two time points - once before intervention (baseline) and once post-intervention (follow-up) - for a total of at least 1,200 exposure measurements. Results will be reported as the mean difference in 24-hour exposure between baseline and follow-up, overall and stratified by household income status.

OTHER OUTCOMES:
Reach: Number and proportion of households reached by implementation strategies | 30 months
  This outcome will assess the reach of the intervention by measuring the number and proportion of households that report exposure to at least one implementation strategy (e.g., direct sales, public sales, stove and electricity subsidies). Data will be collected through a combination of program implementation records and structured household surveys conducted at endline. Results will be reported overall and stratified by household income status.
Adoption: Proportion of recruited implementing organizations that adopt and deliver the implementation strategies as designed | 30 months
  This outcome will assess the adoption of intervention strategies by implementing organizations, including NGOs, government units, sales agents, and local businesses. Adoption is defined as the extent to which each organization delivers the assigned implementation strategies according to protocol. Data will be collected through a combination of program implementation records documenting organizational participation and strategy delivery, and key informant interviews with representatives from each organization to explore fidelity to design, adaptations made, and barriers or facilitators to adoption. The outcome will be reported as the proportion of recruited organizations that adopted and delivered the implementation strategies as originally designed, and findings will be summarized by type of organization.
Implementation: Intervention quality | 30 months
  Proportion of implementers who report that the intervention was delivered with high quality, based on adherence to protocol, clarity of training, perceived effectiveness, and implementation feasibility This outcome will assess the quality of implementation using constructs from the Consolidated Framework for Implementation Research (CFIR) and Proctor's implementation outcomes framework. Data will be collected through key informant interviews with implementing partners and structured implementer surveys. These tools will capture perceptions of implementation processes, adherence to protocol, adaptations made, and barriers or facilitators encountered. Qualitative insights (e.g., from key informant interviews) and quantitative responses (e.g., survey ratings on adherence and quality) will be analyzed together to generate a comprehensive view of implementation quality. Findings will be stratified by type of implementation strategy and by type of stakeholder
Implementation: Intervention fidelity | 30 months
  This outcome will assess the fidelity of implementation using constructs from the Consolidated Framework for Implementation Research (CFIR) and Proctor's implementation outcomes framework. Data will be collected through structured implementer surveys and routine process evaluation tools. These tools will capture adherence to the implementation protocol. Findings will be reported as the proportion of implementation activities delivered as intended, as measured by adherence scores (0-100%), and stratified by type of implementation strategy
Implementation: Intervention acceptability | 30 months
  Proportion of surveyed stakeholders (including household participants and implementers) who report that the intervention was acceptable, based on satisfaction, appropriateness, and ease of implementation or use.
  This outcome will assess the acceptability of implementation using constructs from the Consolidated Framework for Implementation Research (CFIR) and Proctor's implementation outcomes framework. Data will be collected through routine process evaluation tools and household surveys. These tools will capture perceptions of implementation processes adaptations made, and barriers or facilitators encountered. Qualitative insights (e.g., open-ended survey responses, key informant interviews) and quantitative responses (e.g., survey ratings on standardized acceptability scale scores) will be analyzed together to generate a comprehensive view of implementation acceptability. Findings will be stratified by type of implementation strategy and type of stakeholder.
Maintenance: Sustained induction stove use and reduction in biomass stove use at endline. | 30 months
  This outcome will assess the sustainability of induction stove use and the reduction in biomass stove use over time, measured at the endline (18-30 months post-intervention). Data will be collected via structured household surveys that include self-reported frequency of stove use (induction and biomass) and induction stove data loggers. Metrics will include the proportion of households with regular induction stove use and the proportion of households reporting no biomass stove use at endline. These indicators will be reported overall and stratified by household income level.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Freeman, PhD, Principal Investigator — Rollins School of Public Health
Locations (1):
- International Development Enterprises: iDE, Kampong Speu, Kampong Speu Province, Cambodia

IPD SHARING:
Plan to Share IPD: Yes
All de-identified individual participant data collected during the trial. Data sharing will comply with ethical standards and privacy regulations, ensuring individual participant confidentiality is maintained.
  All necessary metadata, tools, and statistical code needed to validate and replicate the findings will be publicly accessible. This includes documentation of the methods used, data collection procedures, and specific parameters for the analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be shared either at the time of publication or at the end of the performance period of the extramural award that produced it, whichever comes first.
Access Criteria: A review committee will evaluate applications. Successful applicants will be required to sign data use agreements outlining the terms and conditions of data access. Data will be made available through a publicly accessible repository, where approved users can access the data, metadata, and any associated documentation